CLINICAL TRIAL: NCT05690867
Title: Comparison of Pressure and Volume Controlled Ventilation in Terms of Mechanical Power in Upper Abdominal Surgery
Brief Title: Pressure Controlled Ventilation Versus Volume Controlled Ventilation in Upper Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Reyhan Nil Kırsan, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2021-2081
Record Dates: First submitted 2022-10-18; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Ventilator Lung
Keywords: mechanical power; volume controlled ventilation; pressure controlled ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): group 1 starts with volume controlled ventilation
  Interventions: Other: Starting with volume controlled ventilation and changing the ventilation mode every 20 minutes
- Group 2 (Other): group 2 starts with pressure controlled ventilation
  Interventions: Other: Starting with pressure controlled ventilation and changing the ventilation mode every 20 minutes

INTERVENTIONS:
Other: Starting with volume controlled ventilation and changing the ventilation mode every 20 minutes — group 1 starts with volume controlled ventilation and we take three consecutive measurements in twenty minutes , after twenty minutes we change the ventilation mode to pressure controlled ventilation after letting washout we take three consecutive measurements at pressure controlled ventilation and we will repeat this protocol during surgery
  Arms: Group 1
Other: Starting with pressure controlled ventilation and changing the ventilation mode every 20 minutes — group 2 starts with pressure controlled ventilation and we take three consecutive measurements in twenty minutes , after twenty minutes we change the ventilation mode to volume controlled ventilation after letting washout we take three consecutive measurements at volume controlled ventilation and we will repeat this protocol during surgery
  Arms: Group 2

SUMMARY:
Comparison of mechanical powers produced at volume controlled and pressure controlled mechanical ventilation

DETAILED DESCRIPTION:
The mechanical power created by mechanical ventilation, as a new concept, can enable to evaluate the effect of different components in the lung.Our aim in this study is to calculate mechanical power in different ventilation modes ( pressure controlled and volume controlled ventilation) and to compare them. To calculate the mechanical powers we will use Van der Meijden's mechanical power formula for pressure controlled ventilation and for volume controlled ventilation we will use Gattinoni's mechanical power formula. In the literature we haven't seen any publication comparing the mechanical power of two commonly used ventilation modes (volume controlled and pressure controlled ventilation)

ELIGIBILITY:
Inclusion Criteria:

* ASA1-2 , >18 years old patients having upper abdominal surgery

Exclusion Criteria:

* chronic obstructive lung disease, interstitial lung disease
* chronic renal failure
* Child-Pugh > 6 liver disease
* Patients who don't give consent
* NYHA > 2 heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
calculation of mechanical power changes in two different ventilation modes | change from at the beginning of surgery till the end of surgery
  mechanical power will be calculated using the Van der Meijden's formula for pressure support ventilation and Gattinoni's formula for volume controlled ventilation and two mechanical powers will be compared

SECONDARY OUTCOMES:
postoperative pulmonary complications | post-operative 7 days
  postoperative pulmonary complication including pneumonia, acute lung injury, respiratory failure requiring reintubation
hospitalisation time | up to 20 days
  up to 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Istanbul University, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Department of Anesthesiology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gattinoni L, Marini JJ, Collino F, Maiolo G, Rapetti F, Tonetti T, Vasques F, Quintel M. The future of mechanical ventilation: lessons from the present and the past. Crit Care. 2017 Jul 12;21(1):183. doi: 10.1186/s13054-017-1750-x. PMID 28701178
- [Background] van der Meijden S, Molenaar M, Somhorst P, Schoe A. Calculating mechanical power for pressure-controlled ventilation. Intensive Care Med. 2019 Oct;45(10):1495-1497. doi: 10.1007/s00134-019-05698-8. Epub 2019 Jul 29. No abstract available. PMID 31359082